CLINICAL TRIAL: NCT05870527
Title: Single-Center Study of Pupillary Dilation During Post-Auricular Vagal Nerve Stimulation
Brief Title: Pupillary Dilation During Post-Auricular Vagal Nerve Stimulation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-00248
Record Dates: First submitted 2023-05-12; First posted 2023-05-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vagal Nerve Stimulation during Cochlear Implantation Surgery (Experimental): Participants undergoing cochlear implantation will receive electrical stimulation during the procedure to stimulate the Arnold's nerve to measure pupil dilation.
  Interventions: Device: Electrical stimulator
- Vagal Nerve Stimulator Implantation (No Intervention): Control cohort undergoing vagal nerve stimulator implantation.

INTERVENTIONS:
Device: Electrical stimulator — Electrical stimulation will be used to stimulate the Arnold's nerve and measure pupil dilation. The electrical stimulator is part of the standard facial nerve monitoring unit that we utilize in cochlear implantation and will be setup prior to surgery in standard fashion. The device allows for constant current stimulation, with stimulus range between 0-30 mA.
  Arms: Vagal Nerve Stimulation during Cochlear Implantation Surgery

SUMMARY:
The research team will evaluate pupillary dilation from vagal nerve stimulation of Arnold's Nerve, a branch of the vagus nerve, during routine cochlear implantation surgery.

DETAILED DESCRIPTION:
The objective of this study is to determine if electrical stimulation of Arnold's Nerve, a branch of the vagus nerve, can result in vagal nerve response through the measurement of pupillary dilation

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing cochlear implantation:

* will be undergoing surgery for a cochlear implant
* is over the age of 18
* is willing to participate in the study

Patients undergoing vagal nerve stimulator implantation:

* will be undergoing implantable vagal nerve stimulation
* is over the age of 18
* is willing to participate in the study

Exclusion Criteria:

Patients undergoing cochlear implantation:

* is under the age of 18
* has history of prior ear surgery, congenital ear malformation, or cochlear implantation
* pregnant or breastfeeding patients cannot undergo the standard-of-care implantation procedures required for participation in the study.
* medical comorbidities resulting in exclusion are guided by the AANS exclusion criteria for VNS and include the following:

  * One vagus nerve
  * Receiving other concurrent forms of brain stimulation
  * Heart arrhythmias or other heart abnormalities
  * Dysautonomias (abnormal functioning of the autonomic nervous system)
  * Lung diseases or disorders (shortness of breath, asthma, etc.)
  * Ulcers (gastric, duodenal, etc.)
  * Vasovagal syncope (fainting)
  * Pre-existing hoarseness

Patients undergoing vagal nerve stimulator implantation:

* is under the age of 18
* has history of prior ear surgery, congenital ear malformation, or cochlear implantation
* pregnant or breastfeeding
* medical comorbidities resulting in exclusion are guided by the AANS exclusion criteria for VNS and include the following:

  * One vagus nerve
  * Receiving other concurrent forms of brain stimulation
  * Heart arrhythmias or other heart abnormalities
  * Dysautonomias (abnormal functioning of the autonomic nervous system)
  * Lung diseases or disorders (shortness of breath, asthma, etc.)
  * Ulcers (gastric, duodenal, etc.)
  * Vasovagal syncope (fainting)
  * Pre-existing hoarseness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pupillary Dilation during Procedure | Day 1 (During procedure - typically 1 hour in duration)
  Pupillary dilation (mm) measured via non-invasive pupillary measurement camera.

CONTACTS AND LOCATIONS:
Overall Officials: J. Thomas Roland Jr., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: justin.cottrell@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to justin.cottrell@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.